CLINICAL TRIAL: NCT06369935
Title: A Real World Study of Equecabtagene Autoleucel in Subjects With Relapsed and Refractory Multiple Myeloma.
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jin Lu, MD, Principal Investigator, Peking University People's Hospital
Other Study IDs: 20240407
Record Dates: First submitted 2024-04-11; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — CT103A chimeric antigen receptor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Equecabtagene Autoleucel — Equecabtagene Autoleucel (CT103A) is a novel fully human BCMA-targeting CAR-T therapy
  Other Names: CT103A

SUMMARY:
This study is a multicenter, observational, single-arm real world study. The purpose of this study is to describe demographic and disease characteristics, treatment patterns, and clinical outcomes in the real-world setting among participants in China with relapsed/refractory multiple myeloma (RRMM) who have been treated with Equecabtagene Autoleucel. This study will use both prospective and retrospective data

DETAILED DESCRIPTION:
Primary endpoint:

Best Overall Response Rate (BOR): The proportion of patients who receive treatment with Ikeolensay injection and have been evaluated by researchers as having the best disease status is strict complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR).

Secondary endpoint:

Progress Free Survival (PFS) rate at 6 months: The probability of patients not experiencing disease progression or death from any cause after receiving treatment with Ikeolensay injection for 6 months; Overall survival (OS) rate at 6 months: the probability of survival of patients after receiving treatment with Ikeolensay injection for 6 months; Time to Response (TTR): The time interval between the patient receiving treatment with Ikeolensay injection and the first recorded time of disease remission; Time to Complete Response (TTCR): The time interval between the patient receiving treatment with Ikeolensay injection and the first recording of complete disease response (CR or sCR); Adverse Event (AE): After receiving treatment with Ikeolensay Injection, researchers consider all adverse events and serious adverse events (SAE) related to Ikeolensay Injection treatment; Hospitalization: After receiving treatment with Ikeolensay injection, the researcher considers any hospitalization related to Ikeolensay injection treatment (including the reason, duration, and outcome of hospitalization); Death: The death of the patient after receiving treatment with Ikeolensay injection, recording the date and cause of death (any reason); Secondary malignant tumors: For any secondary malignant tumors discovered during the monitoring process, researchers can obtain tumor biopsy samples and other necessary samples of tumor tissue according to clinical needs, relevant guiding principles, and product instructions for safety analysis; Quality of life: Evaluate the quality of life using the EQ-5D and EORTCQLQ C30 scoring standards; Medical resource utilization: Collect any medical resource utilization information related to the treatment of patients with Ikeolensay injection (including hospitalization, emergency, outpatient, and new prescription drug usage).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with confirmed relapsed/refractory multiple myeloma;
* Based on clinical practice, the physician decided to administer equecabtagene autoleucel treatment;
* Voluntarily sign the informed consent form approved by the ethics committee.

Exclusion Criteria:

* Patients who are hypersensitive to the active ingredients of the product or any excipients (dimethyl sulfoxide, compound electrolyte injection, human albumin);
* The researcher believes that patients are unable to return for follow-up visits or that it is impossible to complete the study;
* Patients with expected survival less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population of this study was adult patients with relapsed/refractory multiple myeloma who were treated in real world with equecabtagene autoleucel, a commercially available product.
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2026-08-20 (Estimated); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
Best Overall Response Rate， BOR | up to 24 weeks
  Patients treatmented with Equecabtagene Autoleucel, the optimal disease state evaluated by the researcher is strict complete response (sCR),complete response (CR), very good partial response (Very Good Partial Response (VGPR) or partial response (partial response,PR) rate.

SECONDARY OUTCOMES:
PFS rate of 6 month | up to 24 weeks
  Probability of patients not experiencing disease progression or death from any cause 6 months after starting treatment with equecabtagene autoleucel
OS rate of 6 month | up to 24 weeks
  Probability of patient survival 6 months after equecabtagene autoleucel treatment
Time to Response， TTR | up to 24 weeks
  From the time the patient received equecabtagene autoleucel to the first recorded remission of the disease
Time to Complete Response， TTCR | up to 24 weeks
  From the time the patient received equecabtagene autoleucel to the first recorded complete remission of the disease (time interval between CR or sCR)
Adverse Event， AE | up to 24 weeks
  After the patient received treatment with equecabtagene autoleucel, the investigators considered all adverse events and serious adverse events (SAE) related to the treatment with Equecabtagene Autoleucel.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Lu, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No